CLINICAL TRIAL: NCT06886373
Title: Optimizing the Ocular Surface With Systane COMPLETE Pre- and Post-operatively in Patients With Dry Eye Planning for Cataract Surgery: An Extension Study of Optimizing the Ocular Surface With Systane COMPLETE in Patients With Dry Eye Planning for Cataract Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202408096MIND
Record Dates: First submitted 2025-01-23; First posted 2025-03-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Ophthalmology
Keywords: Dry eye; cataract surgery; astigmatism; nano-emulsion; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes; Astigmatism

STUDY DESIGN:
Intervention Model Description: Prospective, double-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systane COMPLETE (Experimental): The experimental group will receive Systane COMPLETE for one month before undergoing the cataract surgery and receive for one month since one week after the surgery.
  Interventions: Drug: Systane Complete
- Control group (No Intervention): The control group will enrolled people who meet the same age and same dry eye syndrome criteria as the experimental group. The control group will not received any intervention.

INTERVENTIONS:
Drug: Systane Complete — Systane COMPLETE is an artificial tears that contain nano-emulsion of mineral oil and phospholipids.
  Arms: Systane COMPLETE

SUMMARY:
Compare the corneal astigmatism data before and after the use of Systane COMPLETE to evaluate its impact on predicting changes in postoperative residual astigmatism, as well as the effects of using or not using Systane COMPLETE on preoperative and postoperative Ocular Surface Disease Index (OSDI) scores and Non-Invasive Tear Break-Up Time (NITBUT).

DETAILED DESCRIPTION:
STUDY OBJECTIVE： Compare the corneal astigmatism data before and after the use of Systane COMPLETE to evaluate its impact on predicting changes in postoperative residual astigmatism.

Compare the effects of using or not using Systane COMPLETE on preoperative and postoperative Ocular Surface Disease Index (OSDI) scores and Non-Invasive Tear Break-Up Time (NITBUT).

Background Cataract surgery is one of the most common and successful ophthalmic surgeries worldwide. However, cataract surgery can induce or exacerbate the severity of dry eye, leading to increased postoperative discomfort for patients. Additionally, undiagnosed preoperative dry eye can affect the accuracy of corneal astigmatism measurements, potentially impacting the astigmatic correction power of toric intraocular lenses used during surgery.

While general moisturizing artificial tears have been shown to significantly reduce postoperative ocular discomfort and tear film instability, it is notable that up to 50% of patients undergoing refractive or cataract surgery exhibit abnormalities in the tear film lipid layer, meeting the diagnostic criteria for meibomian gland dysfunction (MGD).

Given this, the application of lipid-containing nano-emulsion artificial tears before and after cataract surgery presents an unexplored opportunity to address two critical issues: reducing errors in corneal astigmatism measurements and alleviating dry eye symptoms induced by cataract surgery. This remains a topic worthy of investigation, as no existing studies have thoroughly examined these aspects.

Methods This study is an extension of the "Optimizing the Ocular Surface with Systane COMPLETE in Patients with Dry Eye Planning for Cataract Surgery" trial (Research Ethics Committee Approval Number: 202311109MIPD), hereinafter referred to as the OOSSCC trial.

The original OOSSCC trial began recruitment in May 2024 and focuses on analyzing patients with dry eye symptoms scheduled for cataract surgery. The trial evaluates the changes in corneal anterior surface astigmatism measurements, Ocular Surface Disease Index (OSDI) scores, and Non-Invasive Tear Break-Up Time (NITBUT) before and after one month of preoperative treatment with Systane COMPLETE.This trial will extend the study period to one month post-surgery and will be divided into two parts:

Experimental group:

This part extends the use of Systane COMPLETE for participants in the original OOSSCC trial to one month post-surgery. The aim is to compare corneal data before and after using the trial drug to determine which time point provides more accurate predictions of postoperative residual astigmatism. The anticipated results may serve as a reference for preoperative management to reduce corneal astigmatism prediction errors in cataract surgery patients with an OSDI score greater than 12. Additionally, this study aims to assess differences in corneal astigmatism prediction accuracy among patients with varying NITBUT levels.

control group: This part involves recruiting additional cataract patients who meet the same age and dry eye inclusion criteria as the original OOSSCC trial group to serve as a control group. It will compare the effects of using Systane COMPLETE on preoperative dry eye symptoms and postoperative dry eye symptoms. The anticipated results may provide recommendations for managing postoperative dry eye symptoms in cataract surgery patients with an OSDI score greater than 12.

Anticipated Results It is expected that for cataract patients with preoperative dry eye symptoms, particularly those with meibomian gland dysfunction, the study will improve the effectiveness of postoperative astigmatism correction while reducing discomfort caused by dry eye symptoms after surgery.

Hypothesis： Viscous artificial tears have been proven to alter preoperative corneal measurements in patients planning to undergo cataract surgery. This study aims to analyze the impact of lipid-containing nano-emulsion artificial tears on predicting residual astigmatism after cataract surgery.

mpact on Meibomian Gland Dysfunction and Dry Eye Symptoms:Meibomian gland dysfunction is the most common cause of evaporative dry eye. Cataract surgery alters the structure and function of the meibomian glands and reduces the thickness of the tear film lipid layer. However, no studies have yet reported the effectiveness of this type of artificial tear in alleviating dry eye symptoms induced by cataract surgery.

Objectives： Compare the corneal astigmatism data before and after the use of Systane COMPLETE to evaluate its impact on predicting changes in postoperative residual astigmatism.

Compare the effects of using or not using Systane COMPLETE on preoperative and postoperative Ocular Surface Disease Index (OSDI) scores and Non-Invasive Tear Break-Up Time (NITBUT).

Inclusion Criteria (experimental group) Cataract patients who participated in the "Optimizing the Ocular Surface with Systane COMPLETE in Patients with Dry Eye Planning for Cataract Surgery" trial (Research Ethics Committee Approval Number: 202311109MIPD) and did not withdraw from the trial midway.

Exclusion Criteria (experimental group) Patients unwilling to participate in this trial after surgery.

Inclusion Criteria (control group) Cataract patients aged between 20 and 85 years. Patients with normal cognitive function who are able to complete the dry eye questionnaire (with responses recorded by the research team) and are willing to undergo phacoemulsification and intraocular lens implantation under topical anesthesia.

Exclusion Criteria (control group) Unable to answer the questions in the dry eye survey. Ocular trauma or ocular surgery in the planned surgical eye, active ocular infection, and obvious abnormalities in ocular surface or eyelid margins other than MGD cause decreased visual acuity other than cataracts.

Dry eye signs: Corneal Fluorescein Staining CFS (+) to exclude any corneal abnormalities or epithelial defect.

Systemic drug use, including tetracycline derivatives, antihistamines, and isotretinoin.

Using dry eye medication at screening stage.

Sample Size This study plans to enroll a total of 140 participants, with 70 participants in the trial group and 70 in the control group.

ELIGIBILITY:
Inclusion Criteria (Experimental group ): Cataract patients who participated in the "Optimizing the Ocular Surface with Systane COMPLETE in Patients with Dry Eye Planning for Cataract Surgery" trial (Research Ethics Committee Approval Number: 202311109MIPD) and did not withdraw from the trial midway.

Exclusion Criteria (Experimental group ): Patients unwilling to participate in this trial after surgery.

Inclusion Criteria(Control group):

* Cataract patients aged between 20 and 85 years.
* Patients with normal cognitive function who are able to complete the dry eye questionnaire (with - responses recorded by the research team) and are willing to undergo phacoemulsification and intraocular lens implantation under topical anesthesia.

Exclusion Criteria (Control group):

* Unable to answer the questions in the dry eye survey.
* Ocular trauma or ocular surgery in the planned surgical eye, active ocular infection, and obvious abnormalities in ocular surface or eyelid margins other than MGD cause decreased visual acuity other than cataracts.
* Dry eye signs: Corneal Fluorescein Staining CFS (+) to exclude any corneal abnormalities or epithelial defect.
* Systemic drug use, including tetracycline derivatives, antihistamines, and isotretinoin.
* Using dry eye medication at screening stage.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of the keratometry data before and after using Systane COMPLETE | 1-2 months
  The change of the keratometry data is assessed for investigating ocular surface stability after using Systane COMPLETE. The keratometry data is measured using auto-refractor.

SECONDARY OUTCOMES:
The change of the refractive power before and after using Systane COMPLETE | 1-2 months
  The change of the refractive power is assessed for investigating ocular surface stability after using Systane COMPLETE. The refractive power measurement is completed using auto-refractor.
The change of the biometry parameter before and after using Systane COMPLETE | 1-2 months
  The change of the biometry parameters ( ocular length, anterior chamber depth, lens thickness) are assessed for investigating ocular surface stability after using Systane COMPLETE. The biometry parameters is measured using Eyestar 900 (Haag-Streit Diagnostics, Switzerland).
The change of corneal topology map before and after using Systane COMPLETE | 1-2 months
  The change of the corneal topology map is assessed for investigating ocular surface stability after using Systane COMPLETE. The corneal topology map is completed using Pentacam (OCULUS, German), and the corneal optical power is measured.
The change of Ocular Surface Disease Index (OSDI) before and after using Systane COMPLETE | 1-2 months
  Whether Systane COMPLETE relieve dry eye symptoms subjetively is evaluated using the Ocular Surface Disease Index (OSDI) questionnaire. The OSDI questionnaire focuses on three aspects: self-reported eye discomfort, visual function impairment, and environmental triggers. The questionnaire contains 12 items, each rated on a scale from 0 to 4, with a total score ranging from 0 to 100. Higher scores indicate more severe dry eye symptoms. The OSDI questionnaire has high reliability and validity, aiding healthcare professionals in quickly assessing the severity of dry eye, making it suitable for clinical diagnosis and treatment evaluation.
The change of Non-Invasive Tear Break-Up Time (NITBUT) before and after using Systane COMPLETE | 1-2 months
  Whether Systane COMPLETE relieve dry eye symptoms objectively is evaluated using Non-Invasive Tear Break-Up Time (NITBUT). NITBUT is measured using Keratography 5M (K5) to evaluate tear film stability, a key diagnostic indicator for dry eye.

CONTACTS AND LOCATIONS:
Overall Officials: Chiun Ho Hou, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No